CLINICAL TRIAL: NCT00116753
Title: An Open-label Multi-center, Randomized Parallel Group Comparison of Efficacy and Safety of Degarelix Three-Month Depot in Three Different Dosing Regimens in Patients With Prostate Cancer
Brief Title: A Comparative Study of Degarelix Three-month Depot in Three Different Dosing Regimens in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS15
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Degarelix 240@40/240@40 (1,3,6,9) (Active Comparator): 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (40 mg/mL) at months 1, 3, 6 and 9.
  Interventions: Drug: Degarelix
- Degarelix 240@40/240@60(1,3,6,9) (Active Comparator): 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (60 mg/mL) at months 1, 3, 6 and 9.
  Interventions: Drug: Degarelix
- Degarelix 240@40/240@60(1,4,7,10) (Active Comparator): 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (60 mg/mL) at months 1, 4, 7 and 10.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Drug: Degarelix subcutaneous 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (40 mg/mL) at months 1, 3, 6 and 9
  Other Names: FE200486
  Arms: Degarelix 240@40/240@40 (1,3,6,9)
Drug: Degarelix — Drug: Degarelix subcutaneous 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (60 mg/mL) at months 1, 3, 6 and 9
  Other Names: FE200486
  Arms: Degarelix 240@40/240@60(1,3,6,9)
Drug: Degarelix — Drug: Degarelix subcutaneous 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (60 mg/mL) at months 1, 4, 7 and 10
  Other Names: FE200486
  Arms: Degarelix 240@40/240@60(1,4,7,10)

SUMMARY:
The rationale of the study was to evaluate different degarelix dosing regimens for a three-month interval that was to produce and maintain castration in prostate cancer patients through immediate and prolonged testosterone suppression, and to provide confirmatory evidence of the safety of degarelix.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent before any study-related activity is performed. A study-related activity is defined as any procedure that would not have been performed during the normal management of the patient.
* Has a histologically confirmed (Gleason graded) adenocarcinoma of the prostate (all stages) in whom endocrine treatment, except for neoadjuvant hormonal therapy, is indicated. This includes patients with rising PSA after having undergone prostatectomy or radiotherapy with curative intention.
* Is a male patient aged 18 years or over.
* Has a baseline serum testosterone level above the lower limit of normal range, globally defined as >2.2 ng/mL.
* Has an ECOG (Eastern Cooperative Oncology Group) score of 2.
* Has a PSA value of 2 ng/mL.
* Has a life expectancy of at least 13 months.

Exclusion Criteria:

* Has had previous or is currently under hormonal management of prostate cancer (surgical castration or other hormonal manipulation, e.g. GnRH agonists, GnRH antagonists, antiandrogens, oestrogens). However, patients having undergone prostatectomy or radiotherapy with curative intention, neoadjuvant hormonal therapy is accepted for a maximal duration of 6 months. This treatment should have been terminated at least 6 months prior to the Screening Visit.
* Is considered to be a candidate for curative therapy, i.e. radical prostatectomy or radiotherapy within 13 months from Screening Visit.
* Has a history of, or predisposition to, severe hypersensitivity reactions such as severe asthma (defined as a need for daily treatment with inhalation steroids to control the asthma), anaphylactic reactions, or chronic or recurrent urticaria and/or angioedema.
* Has hypersensitivity towards any component of the investigational medicinal product. 5. Has had a cancer disease within the last five years except for prostate cancer and surgically removed basal or squamous cell carcinoma of the skin.
* Has a known or suspected hepatic or symptomatic biliary disease.
* Has elevated serum ALT level above upper level of normal range or serum total bilirubin level above upper level of normal range as measured by the laboratory at the Screening Visit.
* Has other clinically significant laboratory abnormalities, which in the judgment of the investigator would interfere with the patient's participation in this study or evaluation of study results.
* Has a clinically significant disorder (other than prostate cancer) or any other condition, including excessive alcohol or drug abuse, which may interfere with study participation or which may affect the conclusion of the study as judged by the investigator.
* Has a mental incapacity or language barriers precluding adequate understanding or cooperation.
* Has received an investigational drug within the last 28 days preceding Screening Visit or longer if considered by the investigator to possibly influence the outcome of the current study.
* Has previously participated in any degarelix study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (56):
- United States (23):
  - Urology Centers of Alabama, Homewood, Alabama
  - Medical Affiliationed Research Center, Huntsville, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Advanced Urology Medical Center, Anaheim, California
  - Center for Urological Research, La Mesa, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Torrance, California
  - Urology Research Option, Aurora, Colorado
  - South Florida Medical Research, Aventura, Florida
  - RT Services, Inc, Fort Myers, Florida
  - SW Florida Urological Associates, Fort Myers, Florida
  - Regional Urology, Shreveport, Louisiana
  - Mississippi Urology Clinic, Jackson, Mississippi
  - University of Missouri, Urology, Deptof Surgery, Columbia, Missouri
  - Kansas City Urology Care, Kansas City, Missouri
  - Northeast Urology Research, Concord, North Carolina
  - The Urology Center, Greensboro, North Carolina
  - State College Urologic Association, State College, Pennsylvania
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology Association of Northern Texas, Fort Worth, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Seatle Urology Research Centre, Seattle, Washington
- UZ Gasthuisberg Leuven, Leuven, Belgium
- Canada (8):
  - Southern Interior Medical Research Corp, Kelowna, British Columbia
  - Andreou Researce, Surrey, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - The Male/Female Health Centres and Research, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - North Bay Hospital, North Bay, Ontario
  - The Male/Female Health Centres and Research, Oakville, Ontario
  - The Male Health Center, Toronto, Ontario
- Finland (4):
  - Helsinki University Hospital, Maria Hospital, Dept Urology, Helsinki
  - Central Hospital, North Karelian, Dept. of Urology, Joensuu
  - Oulu University Hospital, Department of Surgery Division of Urology, Oys
  - Tampere University Hospital, Dept. of Urology, Tampere
- France (2):
  - Centre Hospitalier Départemental des Oudairies, Chirurgie Urologie, La Roche-sur-Yon
  - Fédération d'Urologie et Néphrologie, Nice
- Germany (2):
  - Gemeinschaftspraxis Dres Effert und Benedic, Aachen
  - Klinik fuer Urologie, Vivantes Klinikum Am Urban, Berlin
- Netherlands (2):
  - Academic Medical Center, Urology, Amsterdam
  - St. Elisabeth Hospital, Tilburg
- Romania (3):
  - Centrul Medical Privat, Arad
  - Clinical Hospital "Prof. Dr. Theodor Burghele", Urology Department, Bucharest
  - University CF Hospital No.2, Urology Clinic, Bucharest
- Russia (5):
  - Andros Clinic, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - Pavlov State Medical University, Outpatient Diagnostic Center affiliated with the Urology Department, Saint Petersburg
  - Pavlov State Medical University, Urology Department, Saint Petersburg
- Serbia and Montenegro (2):
  - Clinical Center of Serbia Institute of Urology and Nephrology, Belgrade
  - Clinical Center Novi Sad, Clinic of Urology Hajduk, Novi Sad
- United Kingdom (4):
  - Ward 10, NHS Forth Valley Acute Operating Division, Falkirk and District Royal Infirmary, Falkirk
  - Mount Vernon Cancer Centre, Marie Curie Research Wing, Middlesex
  - Castle Hill Hospital, Dept. Urology, North Humberside
  - Level 7, Urology Research Unit, Derriford Hospital, Plymouth

RESULTS

PARTICIPANT FLOW:
Groups:
- Degarelix 240@40/240@60 (1,3,6,9): 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (60 mg/mL) at months 1, 3, 6 and 9.
- Degarelix 240@40/240@60 (1,4,7,10): 240 mg (40 mg/mL) initiation dose, maintenance dose 240 mg (60 mg/mL) at months 1, 4, 7 and 10.
Period: Overall Study
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Started | 153 (Randomised.) | 155 | 152
ITT Population | 150 | 150 | 147
Completed | 121 | 125 | 128
Not Completed | 32 | 30 | 24
Not completed — Adverse Event | 16 | 10 | 7
Not completed — Withdrawal by Subject | 11 | 12 | 8
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Did not Fulfil Eligibility Criteria | 1 | 1 | 3
Not completed — Disease Progression | 3 | 4 | 3
Not completed — Abnormal Echocardiogram | 0 | 0 | 1
Not completed — Progressive Parkinson's Disease | 1 | 0 | 0
Not completed — Dosing Error | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10) | Total
Number analyzed (Participants) | 150 | 150 | 147 | 447
Age, Categorical [Count of Participants; unit: Participants] — ITT population. ITT refers to the intent-to-treat population, which includes participants who were both randomized and treated.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 21 | 19 | 20 | 60
    >=65 years | 129 | 131 | 127 | 387
Age Continuous [Median (Full Range); unit: years] — ITT population.
  years | 75 [50 to 86] | 75 [49 to 88] | 75 [50 to 90] | 75 [49 to 90]
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population.
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 150 | 150 | 147 | 447
Race (NIH/OMB) [Count of Participants; unit: Participants] — ITT population.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1 | 2
    Asian | 0 | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    Black or African American | 9 | 15 | 8 | 32
    White | 141 | 131 | 136 | 408
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Curative Intent [Number; unit: Participants] — ITT population. Curative intent refers to radical prostatectomy or radiotherapy.
  Participants
    Yes | 17 | 22 | 17 | 56
    No | 133 | 128 | 130 | 391
Gleason Score [Number; unit: participants] — ITT population. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive. The Gleason scores were missing for two participants.
  participants
    2-4 | 16 | 9 | 15 | 40
    5-6 | 52 | 43 | 61 | 156
    7-10 | 82 | 97 | 70 | 249
Stage of Prostate Cancer [Number; unit: participants] — ITT population. Stage of prostate cancer was classified according to the Tumour, Nodule and Metastatic classification that is a cancer staging system that describes the extent of cancer. T describes the size of the tumor and whether it has invaded nearby tissue, N describes regional lymph nodes that are involved, and M describes distant metastasis.
  participants
    Localized | 56 | 62 | 66 | 184
    Locally advanced | 40 | 31 | 34 | 105
    Metastatic | 28 | 30 | 26 | 84
    Not classifiable | 26 | 27 | 21 | 74
Time Since Prostate Cancer Diagnosis [Mean (Standard Deviation); unit: days] — ITT population.
  days | 465 (1041) | 388 (968) | 346 (738) | 400 (925)
Body Weight [Mean (Standard Deviation); unit: kilogram] — ITT population.
  kilogram | 78.5 (14.6) | 78.4 (13.9) | 77.4 (12.9) | 78.1 (13.8)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — ITT population.
  kilogram per square meter | 25.9 (4.25) | 26.3 (4.42) | 26.0 (4.24) | 26.0 (4.30)
Serum Testosterone Levels [Median (Inter-Quartile Range); unit: nanogram per milliliter] — ITT population.
  nanogram per milliliter | 4.43 [3.19 to 5.74] | 4.00 [3.21 to 5.06] | 4.07 [2.85 to 5.39] | 4.23 [3.08 to 5.45]
Serum Prostate Specific Antigen Levels [Median (Inter-Quartile Range); unit: nanogram per milliliter] — ITT population.
  nanogram per milliliter | 13.8 [6.90 to 48.9] | 16.6 [9.00 to 40.5] | 15.6 [6.20 to 36.2] | 15.6 [7.30 to 40.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Testosterone Level <=0.5 ng/mL From Day 28 Until the End of the Study
Description: Figure in the table give the number of participants with all testosterone values <=0.5 ng/mL from Day 28 to the end of the study.
Time Frame: From Day 28 to 12 or 13 months
Population: Observed Cases in ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Number analyzed (Participants) | 120 | 127 | 129
participants | 94 [69 to 86] | 101 [71 to 87] | 110 [77 to 91]
Statistical Analysis 1: Comparison: Degarelix 240@40/240@40 (1,3,6,9); Test type: Superiority or Other; Percentage of partcipants = 78.3, 96.5% CI 2-sided [69 to 86] — Estimated value is the percentage of participants with all testosterone values from Day 28 to end of study <=0.5 ng/mL. Measure dispersion is the 96.5% two-sided confidence interval which was calculated by the Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 240@40/240@60 (1,3,6,9); Test type: Superiority or Other; Percentage of participants = 79.5, 96.5% CI 2-sided [71 to 87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; Percentage of participants = 85.3, 96.5% CI 2-sided [77 to 91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Degarelix 240@40/240@40 (1,3,6,9) vs Degarelix 240@40/240@60 (1,3,6,9) vs Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; p = 0.3022, Mantel Haenszel
Statistical Analysis 5: Comparison: Degarelix 240@40/240@40 (1,3,6,9) vs Degarelix 240@40/240@60 (1,3,6,9); Test type: Superiority or Other; p = 0.7797, Mantel Haenszel
Statistical Analysis 6: Comparison: Degarelix 240@40/240@40 (1,3,6,9) vs Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; p = 0.1557, Mantel Haenszel
Statistical Analysis 7: Comparison: Degarelix 240@40/240@60 (1,3,6,9) vs Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; p = 0.2208, Mantel Haenszel

2. Secondary Outcome: Number of Participants With Testosterone Level <=0.5 ng/mL After the Dose at Day 28 Until the End of the Study
Description: Figures in the table give the number of participants with all testosterone values <=0.5 ng/mL after the dose at Day 28 to end of study. Thus, the testosterone response after the initial dose is not included in this outcome measure.
Time Frame: From after Day 28 to 12 or 13 months
Population: Observed Cases in ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Number analyzed (Participants) | 119 | 126 | 129
participants | 96 [72 to 88] | 101 [72 to 87] | 111 [78 to 92]
Statistical Analysis 1: Comparison: Degarelix 240@40/240@40 (1,3,6,9); Test type: Superiority or Other; Percentage of participants = 80.7, 96.5% CI 2-sided [72 to 88] — Estimated value is the percentage of participants with all testosterone values from after Day 28 to end of study <=0.5 ng/mL. Measure dispersion is the 96.5% two-sided confidence interval which was calculated by the Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 240@40/240@60 (1,3,6,9); Test type: Superiority or Other; Percentage of participants = 80.2, 96.5% CI 2-sided [72 to 87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; Percentage of participants = 86.0, 96.5% CI 2-sided [78 to 92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Degarelix 240@40/240@40 (1,3,6,9) vs Degarelix 240@40/240@60 (1,3,6,9) vs Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; p = 0.3830, Mantel Haenszel
Statistical Analysis 5: Comparison: Degarelix 240@40/240@40 (1,3,6,9) vs Degarelix 240@40/240@60 (1,3,6,9); Test type: Superiority or Other; p = 0.9587, Mantel Haenszel
Statistical Analysis 6: Comparison: Degarelix 240@40/240@40 (1,3,6,9) vs Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; p = 0.2579, Mantel Haenszel
Statistical Analysis 7: Comparison: Degarelix 240@40/240@60 (1,3,6,9) vs Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; p = 0.2072, Mantel Haenszel

3. Secondary Outcome: Number of Participants With Testosterone <=0.5 ng/mL at Day 28
Description: Figures in the table give number of participants with testosterone <=0.5 ng/mL 28 days after the initial dose of trial medication.
Time Frame: 28 Days
Population: Observed Cases in ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Number analyzed (Participants) | 146 | 146 | 145
participants | 142 [93 to 99] | 143 [94 to 100] | 142 [94 to 100]
Statistical Analysis 1: Comparison: Degarelix 240@40/240@40 (1,3,6,9); Test type: Superiority or Other; Percentage of participants = 97.3, 95% CI 2-sided [93 to 99] — Estimated value is the percentage of participants with testosterone <=0.5 ng/mL at Day 28. Measure dispersion is the 95% two-sided confidence interval which was calculated by the Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 240@40/240@60 (1,3,6,9); Test type: Superiority or Other; Percentage of participants = 97.9, 95% CI 2-sided [94 to 100] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Degarelix 240@40/240@60 (1,4,7,10); Test type: Superiority or Other; Percentage of participants = 97.9, 95% CI 2-sided [94 to 100] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 12 or 13 months
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Number analyzed (Participants) | 150 | 150 | 147
participants
  Abnormal alanine aminotransferase (ALAT) | 60 | 56 | 57
  Abnormal aspartate aminitransferase | 40 | 45 | 50
  Abnormal bilirubin | 4 | 7 | 2
  ALAT >3x upper limit of normal (ULN) | 2 | 2 | 6
  ALAT >3x ULN, bilirubin 1.5x ULN | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Markedly Abnormal Change in Vital Signs and Body Weight as Compared to Baseline
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: 12 or 13 months
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Number analyzed (Participants) | 150 | 150 | 147
participants
  Diastolic blood pressure <=50 and decrease >=15 | 4 | 6 | 2
  Diastolic blood pressure >=105 and increase >=15 | 5 | 7 | 7
  Systolic blood pressure <=90 and decrease >=20 | 1 | 3 | 3
  Systolic blood pressure >=180 and increase >=20 | 5 | 10 | 12
  Heart rate <=50 and decrease >=15 | 6 | 7 | 8
  Heart rate >=120 and increase >=15 | 1 | 2 | 0
  Body weight decrease of >=7 percent | 5 | 4 | 0
  Body weight increase of >=7 percent | 21 | 19 | 17

ADVERSE EVENTS:
Time Frame: 12 or 13 months.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240@40/240@40 (1,3,6,9) | Degarelix 240@40/240@60 (1,3,6,9) | Degarelix 240@40/240@60 (1,4,7,10)
Serious Adverse Events (participants affected / at risk) | 28/150 | 25/150 | 19/147
Other Adverse Events (participants affected / at risk) | 117/150 | 110/150 | 107/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240@40/240@40 (1,3,6,9) (N=150) | Degarelix 240@40/240@60 (1,3,6,9) (N=150) | Degarelix 240@40/240@60 (1,4,7,10) (N=147)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Prostatic specific antigen increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240@40/240@40 (1,3,6,9) (N=150) | Degarelix 240@40/240@60 (1,3,6,9) (N=150) | Degarelix 240@40/240@60 (1,4,7,10) (N=147)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 3 (3) | 6 (6)
Constipation (Gastrointestinal disorders) | 8 (8) | 10 (10) | 5 (9)
Injection site pain (General disorders) | 45 (85) | 31 (68) | 31 (53)
Injection site erythema (General disorders) | 31 (50) | 15 (29) | 17 (25)
Fatigue (General disorders) | 14 (17) | 11 (12) | 11 (12)
Injection site nodule (General disorders) | 10 (16) | 5 (11) | 11 (22)
Injection site swelling (General disorders) | 5 (10) | 13 (24) | 4 (6)
Pyrexia (General disorders) | 12 (18) | 3 (8) | 6 (7)
Injection site induration (General disorders) | 7 (8) | 4 (5) | 9 (14)
Urinary tract infection (Infections and infestations) | 11 (17) | 9 (11) | 9 (11)
Nasopharyngitis (Infections and infestations) | 9 (12) | 11 (15) | 4 (4)
Weight increased (Investigations) | 11 (11) | 9 (10) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (5) | 6 (7) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 6 (6) | 6 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (10) | 7 (10)
Dizziness (Nervous system disorders) | 10 (12) | 12 (14) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (5) | 11 (11) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 7 (7) | 3 (3) | 2 (2)
Hot flush (Vascular disorders) | 57 (60) | 52 (59) | 52 (57)
Hypertension (Vascular disorders) | 4 (5) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.